CLINICAL TRIAL: NCT03025048
Title: PILOT: A Holistic Dietary Intervention for Persons With Spinal Cord Injury
Brief Title: A Holistic Dietary Intervention for Persons With Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: Sunnaas Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Hanne Bjørg Slettahjell, Registered dietitian, MSc, Sunnaas Rehabilitation Hospital
Other Study IDs: 2016/1477-6
Record Dates: First submitted 2017-01-16; First posted 2017-01-19 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: A holistic dietary intervention for persons with spinal cord injury — A lifestyle program over 9 weeks combining individual consultations with a dieatitian and interdiciplinary group sessions

SUMMARY:
People with spinal cord injury are at increased risk for overweight and obesity, type 2 diabetes, cardiovascular disease and decreased quality of life compared With able bodied.

This pilot aims to assess the impact of a nutrition intervention that combines several methods to help people change their lifestyle.

The pilot project combines individual interviews and personal lifestyle goals (diet) with group classes for people with long-standing spinal cord injury.

In addition to nutrition theory and practical exercises for diet-planning, motivational interviewing and mindfullness are incorporated into the course. The course is interdisciplinary, but is led primarily by a dietitian. Data is collected before the course starts and right after the 9-week course ends. The measurements involves self-perceived quality of life, food diary, weight, waist circumference and body composition (measured by BIA and DXA).

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Long-standing Spinal Cord Injury (> 2 years after injury)
* Motivated for lifestyle change

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients With long-standing spinal cord injury (> 2 years after injury)
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Body composition | Short-term: 9 weeks

SECONDARY OUTCOMES:
Diet behaviour | Short-term: 9 weeks

IPD SHARING:
Plan to Share IPD: No